CLINICAL TRIAL: NCT00004810
Title: Phase II Placebo-Controlled Study of 4-Aminosalicylic Acid for Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Vermont (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/12012; UVT-12012
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Ulcerative Colitis
Keywords: gastrointestinal disorders; rare disease; ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative; Gastrointestinal Diseases; Rare Diseases | interventions — Aminosalicylic Acid

INTERVENTIONS:
Drug: -aminosalicylic acid

SUMMARY:
OBJECTIVES:

I. Assess the safety and efficacy of 4-aminosalicylic acid in patients with mildly to moderately severe ulcerative colitis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized study. Patients are stratified by extent of disease.

Patients are randomly assigned to oral 4-aminosalicylic acid (4-ASA) or placebo administered daily for 6 weeks. Optional 4-ASA is available to all patients for up to 1 year.

Concurrent therapy with low-dose sulfasalazine, prednisone, or equivalent is allowed.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

* Mildly to moderately severe ulcerative colitis
* Patient age: 18 to 80

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 1996-06

CONTACTS AND LOCATIONS:
Overall Officials: Warren L. Beeken, Study Chair — University of Vermont

REFERENCES:
- [Background] Beeken W, Howard D, Bigelow J, Trainer T, Roy M, Thayer W, Wild G. Controlled trial of 4-ASA in ulcerative colitis. Dig Dis Sci. 1997 Feb;42(2):354-8. doi: 10.1023/a:1018874120749. PMID 9052519